CLINICAL TRIAL: NCT00130130
Title: Testing the Effects of an Algorithm for Neuropathic Pain on Patient and System Outcomes
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D 0403; ONS
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The overall purpose of this project is to improve nurse skills regarding neuropathic pain (NP) assessment, treatment and referral practices through implementation of an evidence-based algorithm and to improve selected patient outcomes as a result of algorithm use.

DETAILED DESCRIPTION:
Neuropathic pain (NP) is defined as pain that arises from injury, disease or dysfunction of the central or peripheral nervous system. For the patient focused phase of the project NP treatment will be guided via the Peripheral Neuropathy Treatment Algorithm. Patients will receive algorithm-specific treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients experiencing NP from a variety of causes
* NP Visual Analogue Scale (VAS) score equal to or > 4 with 12 week estimated duration
* Karnofsky Performance Status (KPS) 60% or greater
* Age greater than 18

Exclusion Criteria:

* Patients undergoing anticancer or invasive pain procedures specifically intended to palliate NP are ineligible

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients experiencing NP from a variety of causes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To implement an evidence based screening, assessment, treatment, and referral guideline for hematology/oncology patients with NP receiving care | outcome measures will consist of the NPVAS, and a PPCPS adapted rom the original project. Adequate satisfaction will be defined as 25% or mor of all patients reporting being very or completely satisfied as measured by PPCPS

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Lavoie-Smith, ARNP, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States